CLINICAL TRIAL: NCT06650241
Title: A Clinical Comparative Study of Different Methods for Correcting Lower Lip Sucking Habits in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Guo Xueqiang, phD, Qingdao University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QFELL-YJ-2016-66
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Oral Habits
Keywords: preschool children, Oral Health-Related Quality of Life (OHRQoL), Early Childhood Oral Health Impact Scale (ECOHIS),
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- Behavioral therapy (Experimental): Behavioral Therapy Group: Children were rewarded with their favorite candy or toys as positive reinforcement when they refrained from sucking their lower lip. When they exhibited lip-sucking behavior, corresponding punishments were applied (e.g., being prohibited from watching cartoons for 1 hour or from playing with toys) as negative reinforcement. At night, bitter nail polish or substances with unpleasant smells were applied to the lower lip as aversive stimuli. Patients attended follow-up appointments monthly.
  Interventions: Other: Behavioral therapy
- Maxillary lip bumper appliance (Experimental): Lip Bumper Therapy Group: The treatment involved placing arrow-shaped clasps and interproximal hooks on the maxillary molars, with a double-curved labial bow positioned on the labial side of the upper anterior teeth. A lip bumper wire was soldered at the position of the maxillary central incisors. The lip bumper wire should reach the mandibular vestibular groove to support the lower lip without obstructing the natural labial adjustment of the lower anterior teeth. Patients were required to wear the appliance at all times except during meals and oral hygiene activities. Monthly follow-up appointments were conducted, during which the double-curved labial bow could be adjusted to retract the upper anterior teeth.
  Interventions: Other: Lip Bumper Therapy
- Twin-block (Experimental): Modified Twin-Block Therapy Group: Initially, occlusal reconstruction was performed, with the combined forward movement of the mandible and vertical dimension being less than 10 mm. The standard criteria were an incisal edge-to-edge bite of the upper and lower anterior teeth, with the vertical opening in the posterior region exceeding the resting occlusal gap by 2-3 mm. Patients were required to wear the appliance at all times except during meals and oral hygiene activities. Monthly follow-up appointments included progressive grinding of the maxillary occlusal pads. If discrepancies in arch width occurred, expansion therapy was implemented.
  Interventions: Other: Modified Twin-Block Therapy

INTERVENTIONS:
Other: Behavioral therapy
  Arms: Behavioral therapy
Other: Lip Bumper Therapy
  Arms: Maxillary lip bumper appliance
Other: Modified Twin-Block Therapy
  Arms: Twin-block

SUMMARY:
Comparison of the Effectiveness of Behavioral Therapy, Maxillary Lip Bumper Appliance, and Twin-Block Appliance in Correcting Lower Lip Sucking Habits in Children

DETAILED DESCRIPTION:
Intervention Methods Behavioral Therapy Group: Children were rewarded with their favorite candy or toys as positive reinforcement when they refrained from sucking their lower lip. When they exhibited lip-sucking behavior, corresponding punishments were applied (e.g., being prohibited from watching cartoons for 1 hour or from playing with toys) as negative reinforcement. At night, bitter nail polish or substances with unpleasant smells were applied to the lower lip as aversive stimuli. Patients attended follow-up appointments monthly.

**Lip Bumper Therapy Group:** The treatment involved placing arrow-shaped clasps and interproximal hooks on the maxillary molars, with a double-curved labial bow positioned on the labial side of the upper anterior teeth. A lip bumper wire was soldered at the position of the maxillary central incisors. The lip bumper wire should reach the mandibular vestibular groove to support the lower lip without obstructing the natural labial adjustment of the lower anterior teeth. Patients were required to wear the appliance at all times except during meals and oral hygiene activities. Monthly follow-up appointments were conducted, during which the double-curved labial bow could be adjusted to retract the upper anterior teeth.

Modified Twin-Block Therapy Group: Initially, occlusal reconstruction was performed, with the combined forward movement of the mandible and vertical dimension being less than 10 mm. The standard criteria were an incisal edge-to-edge bite of the upper and lower anterior teeth, with the vertical opening in the posterior region exceeding the resting occlusal gap by 2-3 mm. Patients were required to wear the appliance at all times except during meals and oral hygiene activities. Monthly follow-up appointments included progressive grinding of the maxillary occlusal pads. If discrepancies in arch width occurred, expansion therapy was implemented.

Evaluation of Therapeutic Efficacy

All children were assessed for the following indicators after 6 months of treatment:

1. Comparison of Lip-Sucking Habit Improvement: The outcome of lip-sucking habit correction was compared among the groups. Treatment was considered successful if the lip-sucking habit was completely corrected, malocclusion was improved, and parents were satisfied. It was considered unsuccessful if there was no significant improvement in the lip-sucking habit and parents were dissatisfied. Success rate = (Number of successful cases / Total number of cases) × 100%.
2. Comparison of Oral Examination and Model Analysis Indicators:** Oral examinations and oral model preparation were conducted before treatment (T0) and one month after the end of treatment (T2). Changes in the overjet of the anterior teeth were measured using a vernier caliper.
3. Comparison of Cephalometric Measurements:Lateral cephalometric radiographs were taken before treatment (T0) and one month after the end of treatment (T2). SNA, SNB, ANB, U1-SN, and L1-MP angles were measured using Dolphin software (Version 11.8, Dolphin Imaging and Management Solutions, CA, USA).
4. Assessment of Oral Health-Related Quality of Life (OHRQoL) using the ECOHIS Questionnaire:The Chinese version of the Early Childhood Oral Health Impact Scale (ECOHIS) was used to assess the impact of lip-sucking habits and orthodontic treatment on children's OHRQoL. Parents completed the ECOHIS questionnaire before treatment (T0), after 1 month of treatment (T1), and 1 month after the end of treatment (T2). The questionnaire includes 13 items, covering the *Child Impact Section* (CIS) which assesses the impact on the child's symptoms, functions, psychology, and social interactions, as well as the *Family Impact Section* (FIS), which assesses the impact on parental distress and family function. Each item is rated on a scale of 0-5: never (0), hardly ever (1), occasionally (2), often (3), very often (4), don't know (5). The total ECOHIS score is calculated by summing the response codes from both CIS and FIS sections. The score ranges from 0 to 65, with higher scores indicating a greater negative impact on children's OHRQoL. The questionnaire was considered invalid if there were more than two "don't know" responses in the CIS or one in the FIS, and another child was selected for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children aged 3-6 years,
* Habit of lower lip sucking,
* No anterior crossbite or open bite,
* Missing no more than 2 incisors in a single jaw,
* No other systemic diseases,
* The child's family has a certain level of reading and comprehension ability, can effectively understand the questionnaire content, and is willing to sign the informed consent form.

Exclusion Criteria:

* Prior orthodontic treatment;
* Tooth extraction;
* Mini-implant usage;
* Chronic rhinitis, tonsil hypertrophy and other upper airway diseases.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
overjet | 6 months
  Overjet refers to the horizontal distance between the front edge of the upper front teeth (maxillary incisors) and the front edge of the lower front teeth (mandibular incisors). In a normal alignment, the upper front teeth slightly overlap the lower front teeth, but when this overlap is excessive, it results in a noticeable overjet.
  From a side view, overjet is measured as the horizontal distance between the upper and lower front teeth, typically in millimeters. A normal overjet is usually around 2-3 millimeters. If the distance is greater than this, it is considered abnormal. A large overjet can lead to issues with bite alignment, aesthetics, and function, such as difficulties with eating or speaking, and increased vulnerability to trauma.
ANB | 6 months
  ANB is an angle measurement used in orthodontics and cephalometrics to evaluate the relative position of the maxilla (upper jaw) to the mandible (lower jaw). It is derived from the difference between the SNA and SNB angles:
  S (Sella): The center of the sella turcica. N (Nasion): The junction of the frontal bone and nasal bones at the bridge of the nose.
  A (Point A): A point on the deepest curve of the maxillary alveolar bone. B (Point B): A point on the deepest curve of the mandibular alveolar bone. The ANB angle is calculated as SNA - SNB, providing an assessment of the relationship between the upper and lower jaws. It is typically used to diagnose skeletal discrepancies, such as Class I, Class II, or Class III jaw relationships.
ECOHIS | 6 months
  ECOHIS, or the Early Childhood Oral Health Impact Scale, is a questionnaire designed to assess the impact of oral health problems and dental treatments on the quality of life of young children and their families. It is specifically aimed at children aged 0 to 5 years and evaluates the broader effects of oral health issues beyond just clinical symptoms.
  The ECOHIS is valuable in research and clinical practice as it helps to understand the broader impact of oral health issues, guiding treatment planning and interventions aimed at improving not only the clinical condition but also the overall well-being of young children and their families.

SECONDARY OUTCOMES:
SNB | 6 months
  SNB is an angle measurement used in orthodontics and cephalometrics to assess the position of the mandible (lower jaw) relative to the cranial base. It is measured using three reference points:
  S (Sella): The center of the sella turcica, a cavity in the sphenoid bone that houses the pituitary gland.
  N (Nasion): The point where the frontal bone and the nasal bones meet, located at the bridge of the nose.
  B (Point B): A point on the deepest curvature of the mandibular alveolar process, which is the bone that holds the lower teeth.
  The SNB angle helps determine whether the mandible is positioned normally, or if it is too far forward (protrusive) or too far back (retrusive) relative to the cranial base. A typical SNB value is around 80 degrees. Higher values indicate mandibular protrusion, while lower values suggest mandibular retrusion. This measurement is essential for diagnosing skeletal discrepancies and planning orthodontic treatments that address the alignment of the jaws.
SNA | 6 months
  SNA is an angle measurement used in orthodontics and cephalometrics to assess the position of the maxilla (upper jaw) relative to the cranial base. It is measured by evaluating the angle between three points:
  S (Sella): The center of the sella turcica, a cavity in the sphenoid bone that houses the pituitary gland.
  N (Nasion): The point where the frontal bone and the nasal bones meet, located at the bridge of the nose.
  A (Point A): A point on the deepest curvature of the maxillary alveolar process, which is the bone that holds the upper teeth.
  The SNA angle helps determine whether the maxilla is positioned normally, or if it is too far forward (protrusive) or too far back (retrusive) relative to the cranial base. A typical SNA value is around 82 degrees. Higher values suggest maxillary protrusion, while lower values indicate maxillary retrusion. This measurement is crucial in diagnosing and planning treatments for orthodontic and skeletal alignment issues.
U1SN | 6 months
  U1SN is an orthodontic cephalometric measurement that assesses the angulation of the upper front teeth (upper incisors) relative to the cranial base. It helps determine the inclination of the maxillary incisors and is measured as the angle between two lines:
  U1 (Upper Incisor Line): A line that runs through the long axis of the upper central incisor.
  SN (Sella-Nasion Line): A line that connects the Sella (S) point to the Nasion (N) point, representing the base of the skull.
  The U1SN angle indicates the degree of forward or backward tilt of the upper incisors. Typical values range between 102 to 110 degrees.
L1MP | 6 months
  L1MP is a cephalometric measurement used in orthodontics to assess the inclination of the lower front teeth (lower incisors) relative to the mandibular plane. It helps to determine the angulation of the lower incisors and is measured as the angle between two lines:
  L1 (Lower Incisor Line): A line drawn through the long axis of the lower central incisor.
  MP (Mandibular Plane): A line that typically runs from the Menton (the lowest point on the chin) to the Gonion (the angle of the jaw).
  The L1MP angle indicates the degree of forward or backward tilt of the lower incisors. Normal values for this angle are usually around 90 to 95 degrees.

IPD SHARING:
Plan to Share IPD: No